CLINICAL TRIAL: NCT04877795
Title: Predictive Value of Copeptin and Heart-Type Fatty Acid Binding Protein in Cardiac Surgery - A Multicenter Prospective Cohort Study
Brief Title: Copeptin and HFABP in Cardiac Surgery
Acronym: PRACTICE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: V1.0
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Coronary Artery Disease; Valvular Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Surgery: Adult Patients undergoing elective on-pump cardiac surgery (i.e. Coronary artery bypass graft surgery (CABG) and/or valvular surgery)
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — Blood will be sampled from enrolled patients and analyzed for levels of troponin, copeptin and heart-type fatty acid binding protein (HFABP).

SUMMARY:
In-hospital mortality after cardiac surgery ranges from 2-6%. Many patients suffer from major adverse cardiovascular events (MACE) which results in impaired disability-free survival. Troponin plays the central role in identifying MACE. However, interpretation after cardiac surgery is difficult due to ischemia-reperfusion-injury and direct surgical trauma. While the 4th universal definition of type 5 myocardial infarction uses the 10 x ULN as cut-off, >90% of patients after on-pump procedures exceed this cut-off. Clinical consequences are unclear. The dynamic of Copeptin and Heart-type fatty acid binding protein (H-FABP) concentrations starts very early, i.e. several hours before Troponin. The investigators plan a prospective multicenter cohort study to evaluate 1) the independent association between Copeptin and H-FABP with disability -free survival and MACE after cardiac surgery; 2) the predictive gain of their addition to the Euroscore II; 3) the independent association between H-FABP and acute kidney injury.

DETAILED DESCRIPTION:
The initial patient visit will take place after screening of patients and eligibility assessment and no later than on the day before surgery (day -1). After provision of patient information and written informed consent, baseline data will be extracted from clinical source documents. Blood will be sampled prior to induction (Troponin), upon arrival in the intensive care unit (Troponin, HFABP and Copeptin), and on postoperative day 1 and 2 (Troponin). Sampling will occur as far as possible concurrently to clinically indicated blood samples. Blood samples will be analyzed in a certified laboratory.

All patients will be contacted after 30 days and 12 months by E-Mail, postal mail and/or phone call to obtain for the 12-item WHODAS 2 and information on potential events.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years of age)
* Elective surgery
* On-pump cardiac surgery (CABG and/or valvular surgery)

Exclusion Criteria:

* Heart transplantation (HTX)
* ACS at presentation (< 14 days)
* Emergency surgery
* Preoperative inotropic or mechanical circulatory support
* Left or right ventricular assist device implantation
* Unwilling or unable to provide consent
* Inability to follow the procedures of the study, e.g. due to language barriers, psychiatric disorders, dementia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective on-pump cardiac surgery (i.e. CABG and/or valvular surgery).
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Disability-free survival | 1 years after surgery
  Disability is defined as a persistent (at least 6 months) impairment in health status, as measured by the 12-item WHODAS 2.0 score, of at least 24 points when using response scores of 1-5 for each item, reflecting a disability level of at least 25% and being the threshold point between 'disabled' and 'not disabled' as per WHO guidelines.

SECONDARY OUTCOMES:
Days alive and out of hospital | At 30 days and 12 months after surgery
  Patient-centered outcome to measure morbidity and mortality after surgery
Major adverse cardiovascular events (MACE) | At 30 days and 12 months after surgery
  Defined as non-fatal cardiac arrest, acute myocardial infarction, congestive heart failure or transfer to a higher unit of care, atrial fibrillation or stroke
All cause mortality | At 30 days and 12 months after surgery
  Evaluate mortality after cardiac surgery
Length of ICU-stay | At 30 days
  To observe the length and/or readmission rate of intensive care unit stay
Acute kidney injury (AKI) | At 30 days
  As defined by the three-stage KDIGO (Kidney Disease: Improving Global Outcome) classification of severity

CONTACTS AND LOCATIONS:
Locations (1):
- Heinrich-Heine-Universität, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
Data will be entered into a secure on-line database documenting the time and individual entering the data. Data will be collected directly from source documents into the eCRF. A copy of the original source documents will be stored within a locked cabinet/office accessible to authorized personnel only. An identifiable patient data page reporting the assigned patient identification code will be stored separately also in a locked cabinet/office (accessible to authorized personnel only) in order to record in-hospital outcomes, conduct follow-up, supply missing data points, and to allow potential monitoring visits by regulatory authorities. All collected data will be archived for a period of 15 years.
  The secure database run by the clinical trials unit of the University Hospital Duesseldorf allows for data entry accountability and high security standards.

REFERENCES:
- [Derived] Kirkopoulos A, Salehi I, M'Pembele R, Maddison P, Stroda A, Tenge T, Donaldson D, Huhn R, Kindgen-Milles D, Haddad A, Brands J, Dubler S, Brenner T, Berger MM, Lurati Buse G, Roth S. Predictive value of early postoperative copeptin after cardiac surgery: A two-centre prospective cohort study. Eur J Anaesthesiol. 2025 Nov 1;42(11):1017-1024. doi: 10.1097/EJA.0000000000002251. Epub 2025 Aug 1. PMID 40755220